CLINICAL TRIAL: NCT05181761
Title: Do Healthcare Personnel Wearing Non-chipped, Gel Nail Polish Harbor Increased Nail Bacterial Counts in Comparison to Healthcare Personnel Without Nail Polish
Brief Title: Prospective Nail Polish Study
Acronym: Nail Polish
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2021-0810
Record Dates: First submitted 2021-12-20; First posted 2022-01-06 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Bacterial Growth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Left Hand with gel polish (Experimental): The participants will receive gel nail polish on their left hand. The right hand will remain natural (no gel polish)
  Interventions: Other: Gel Polish
- Right Hand with gel polish (Experimental): The participants will receive gel nail polish on their right hand. The left hand will remain natural (no gel polish).
  Interventions: Other: Gel Polish

INTERVENTIONS:
Other: Gel Polish — One hand of a subject with receive nail polish to compare bacterial growth between hands with gel nail polish to those without.

SUMMARY:
This is an randomized, prospective study utilizing volunteers from the anesthesia department at Geisinger Medical Center (GMC). Subjects' hands will be randomized 1:1 using statistical software to determine which hand will receive the gel polish using proportional stratified random sampling. The glove juice method will be used to measure hand bacterial counts to determine whether or not hands with nail polish harbor more bacteria than hands without polish. In addition, all subjects will fill out an employee satisfaction survey related to their satisfaction at work at the beginning of the study as well as at the end of the study.

DETAILED DESCRIPTION:
The study is recruiting Geisinger employees who are 18 years old that work as Anesthesiologists, Anesthesia resident physicians, Certified Registered Nurse Anesthetists (CRNA) in the anesthesia department involved in direct patient care. The study duration will be one month (30 days). On day zero, participants' baseline hand bacteria counts will be measured for each hand via the glove juice method. Subsequently, after participants' hands have been randomized into the painted and unpainted groups, they will receive a manicure on either their left or right hand. In other words, if a patient's left hand is randomized into the painted group, then that hand will be painted, and the right hand will be left unpainted, and vice versa. All participants will then be seen on days 1, 7, 14, 21, and 28 to have both hand's bacterial counts measured.

On study day zero, all subjects will meet at a designated Geisinger Medical Center location and will be asked to fill out a work satisfaction survey. Then, before the subjects' hands are randomized into painted and unpainted groups, each of their hands' baseline bacteria counts will be measured using the glove juice method.

Measuring hand bacteria counts with the glove juice method:

Prior to performing the glove juice method to obtain hand bacteria counts, participants will be asked to wash their hands with soap and water. Participants will then place their hands into regular, non-sterile gloves. The premade broth for the glove juice method will then be placed into both gloves. The study group administrators will then place an elastic around both subject's wrists so that the juice does not spill out of the gloves. Hands will be gently massaged for one minute. Then, for each gloved hand, a pipet will remove some of the juice and this will be sent to the laboratory to determine the juice bacterial counts (log10CFU). The bacterial counts will be recorded on that particular subject's Bacterial count form and later entered into REDCap. After recording the specimens will be discarded.

All subjects will then return on days 1, 7, 14, 21, and 28. The study administrators will directly record whether or not there are any chips on the nails of the hands in the nail polish group and record their findings on the subject's bacterial count sheet. All subjects will have the glove juice method previously described performed again. Juice specimens obtained on each date will be sent to the laboratory and bacterial counts recorded on the bacterial count sheet and later entered into REDCap.

ELIGIBILITY:
Inclusion Criteria:

* Geisinger employee
* ≥18 years of age
* Able and willing to provide consent
* Works as a Anesthesiologists, Anesthesia resident physicians or Certified Registered Nurse Anesthetists (CRNA))

Exclusion Criteria:

* Hospital employees in the anesthesia department that are not involved in direct patient contact (Anesthesia Technicians).
* Hospital employees that are under 18 years of age

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-09-11 (Actual); Primary Completion 2022-11-21 (Actual); Study Completion 2023-03-24 (Actual)

PRIMARY OUTCOMES:
Rate of hand bacterial growth in natural nails and polished nails | 6 months
  To compare the rate of growth of bacteria found on the hands with natural nails versus nails with gel polish.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Hoffman, MD, Principal Investigator — Geisinger Physician
Locations (1):
- Geisinger, Danville, Pennsylvania, United States